CLINICAL TRIAL: NCT04908748
Title: The Efficacy and Safety of an Esflurbiprofen Hydrogel Patch vs. Placebo in the Local Symptomatic and Short-term Treatment of Pain in Acute Strains, Sprains or Bruises of the Extremities Following Blunt Trauma, e.g. Sports Injuries.
Brief Title: Efficacy and Safety of Esflurbiprofen Hydrogel Patch in the Treatment of Local Acute Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: ClinSearch (Other); CRM Biometrics GmbH (Industry); Clinigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TK-254R-0201
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Soft Tissue Injuries; Contusions; Strains; Sprains; Bruises
Keywords: Blunt Trauma
MeSH Terms: conditions — Soft Tissue Injuries; Contusions; Sprains and Strains; Wounds, Nonpenetrating

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind, multi-center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Packages of Investigative Medicinal product will be non-distinguishable to patients, study site staff and monitors.
  Randomization data are kept strictly confidential, accessible only to authorized persons, until the time of unblinding the identity of the treatments will be concealed by the use of study drugs that are all identical in packaging, labeling, schedule of administration, appearance and odor.
  Unblinding will only occur in the case of patient emergencies and at the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): Esflurbiprofen Hydrogel Patch containing 165 mg Esflurbiprofen
  Interventions: Drug: Esflurbiprofen Hydrogel Patch
- Control Drug (Placebo Comparator): Placebo patch that does not contain the active ingredient but is otherwise indistinguishable from the investigational drug Esflurbiprofen Hydrogel Patch
  Interventions: Drug: Esflurbiprofen Hydrogel Patch

INTERVENTIONS:
Drug: Esflurbiprofen Hydrogel Patch — Esflurbiprofen is a cyclooxygenase (COX) inhibitor

SUMMARY:
Objective of this study is:

to determine efficacy and safety of a Esflurbiprofen Hydrogel Patch compared to placebo in patients with acute strains, sprains or bruises of the extremities following blunt trauma, e.g. sports injuries.

to demonstrate that the Esflurbiprofen Hydrogel Patch is superior to placebo, and that the patch has acceptable local tolerability.

DETAILED DESCRIPTION:
Study Design Randomized (1:1) (stratified by center and 2 subgroups), controlled, double-blind, multi-centric study in parallel groups. Patient Population/Sample size/Study Sites

The clinical trial population will consist of male or female patients, 18 - 60 years suffering from acute; strains, sprains or bruises of the extremities following blunt trauma, and meeting all clinical trial entry criteria.

200 patients will be enrolled (assumes a drop-out-rate of ≤10%).

The study will be performed in Germany in 3 sites

ELIGIBILITY:
Inclusion criteria

1. acute sports-related soft-tissue injury/contusion (strains, sprains, bruises) of the upper or lower limb
2. location of injury such that pain-on-movement (POM) is elicited on by specified exercises
3. enrollment within 6 hours of the injury
4. baseline VAS score for POM of injured extremity > 50 mm on a 100 mm VAS
5. size of injury, as assessed by investigator, ≥ 25 cm2 and ≤ 120 cm2
6. adult male or female patients
7. age 18 to 60 years
8. having given written informed consent
9. satisfactory health as determined by the Investigator based on medical history and physical examination.

Exclusion criteria

1. significant concomitant injury in association with the index acute sports-related soft- tissue injury/contusion; e.g. fracture, nerve injury, ligament disruption, tear of muscle or cartilage, or open wound
2. excessively hairy skin at application site, cutting the hair in the injured site prior to patch application will qualify for inclusion
3. current skin disorder or shaving hair at application site
4. history of excessive sweating/hyperhidrosis inclusive of application site
5. intake of NSAIDs or analgesics within 36 hours, opioids within 7 days, or corticosteroids within 60 days of inclusion in the study
6. intake of long-acting NSAIDs or application of topical medication since the injury (RICE allowed)
7. participation in a clinical study within 30 days before inclusion in the study or concomitantly
8. drug or alcohol abuse in the opinion of the investigator
9. Pregnant and lactating women
10. Women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) who are not using an acceptable method of contraception defined as:

    * Surgical sterilization
    * Hormonal contraception
    * Intra Uterine Device
    * Double barrier method
    * Total abstinence throughout the study at the discretion of the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Aoki, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (1):
- Deutsche Sporthochschule Köln Institut für Kreislaufforschung und Sportmedizin, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Arm | Control Drug
Started | 98 | 102
Completed | 98 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Control Drug | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (11.0) | 34.3 (10.8) | 33.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 47 | 102
  Male | 43 | 55 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 60 | 64 | 124
  Unknown or Not Reported | 37 | 36 | 73
Region of Enrollment [Number; unit: participants]
  Germany | 98 | 102 | 200
Type of injury [Count of Participants; unit: Participants]
  Contusions | 73 | 72 | 145
  Sprains＆Strains | 25 | 30 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain-on-movement (POM) Compared to Baseline
Description: Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: Change from baseline to Visit 5 (72 hours after initiating treatment)
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
units on a scale | -50.7 (11.1) | -21.6 (11.9)
Statistical Analysis 1: Comparison: Active Arm vs Control Drug; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -29.1, 95% CI 2-sided [-32.2 to -26.0]

2. Secondary Outcome: Pain-on-movement (POM) on VAS
Description: Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: Baseline and 12, 24, 48, 72, 96, 168 hours after initiating treatment
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
units on a scale
  Baseline | 69.9 (7.6) | 70.1 (8.3)
  12 hour | 61.1 (10.3) | 66.4 (8.4)
  24 hour | 48.8 (12.2) | 62.8 (10.4)
  48 hour | 33.3 (11.9) | 56.6 (12.0)
  72 hour | 19.2 (9.7) | 48.5 (14.9)
  96 hour | 9.2 (8.3) | 37.3 (16.7)
  168 hour | 2.1 (4.4) | 19.4 (17.4)

3. Secondary Outcome: Area-under-the-curve for POM on VAS
Description: Area-under-the-curve (AUC) over time during first 12, 24, 48, 72, 96 and 168 hours for Pain on movement (POM) measured using a VAS Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: Baseline and 12, 24, 48, 72, 96, 168 hours after initiating treatment
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Mean (Standard Deviation); unit: AUC of POM VAS pain (mm* h)
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
AUC of POM VAS pain (mm* h)
  0-12 h | 814.9 (107.0) | 842.9 (109.3)
  0-24 h | 1424.5 (210.3) | 1556.3 (182.6)
  0-48 h | 2397.3 (448.7) | 2970.3 (415.3)
  0-72 h | 3026.1 (655.8) | 4242.4 (730.3)
  0-96 h | 3367.6 (818.9) | 5300.7 (1166.8)
  0-168 h | 3771.4 (1149.6) | 7285.7 (1952.1)

4. Secondary Outcome: Pain-at-rest on VAS
Description: Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: Baseline and 12, 24, 48, 72, 96, 168 hours after initiating treatment
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
units on a scale
  Baseline | 17.9 (5.9) | 17.0 (7.7)
  12 h | 14.7 (6.1) | 15.2 (6.4)
  24 h | 11.2 (5.4) | 13.5 (6.2)
  48 h | 7.5 (4.6) | 11.5 (6.2)
  72 h | 4.1 (3.4) | 9.2 (5.5)
  96 h | 2.0 (2.7) | 6.5 (5.4)
  168 h | 0.5 (1.5) | 3.7 (4.4)

5. Secondary Outcome: Time to Meaningful and Optimal Reduction
Description: The time taken to achieve a meaningful (30 %) and optimal (50 %) reduction of pain measured on the VAS for POM Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: Baseline and 12, 24, 48, 72, 96, 168 (192) hours after initiating treatment
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants
  Time to meaningful reduction of pain (h) (30% or more): < 12 | 8 | 1
  Time to meaningful reduction of pain (h) (30% or more): 12-24 | 41 | 3
  Time to meaningful reduction of pain (h) (30% or more): 24-48 | 42 | 10
  Time to meaningful reduction of pain (h) (30% or more): 48-72 | 7 | 33
  Time to meaningful reduction of pain (h) (30% or more): 72-96 | 0 | 35
  Time to meaningful reduction of pain (h) (30% or more): 96-192 | 0 | 15
  Time to meaningful reduction of pain (h) (30% or more): Not achieved | 0 | 5
  Time to optimal reduction of pain (h) (50 % or more): < 12 | 2 | 0
  Time to optimal reduction of pain (h) (50 % or more): 12-24 | 4 | 1
  Time to optimal reduction of pain (h) (50 % or more): 24-48 | 51 | 1
  Time to optimal reduction of pain (h) (50 % or more): 48-72 | 36 | 13
  Time to optimal reduction of pain (h) (50 % or more): 72-96 | 5 | 26
  Time to optimal reduction of pain (h) (50 % or more): 96-192 | 0 | 42
  Time to optimal reduction of pain (h) (50 % or more): Not achieved | 0 | 19

6. Secondary Outcome: Time to Complete Resolution of Pain
Description: Time to complete resolution of pain, i. e. reaching a POM VAS value of 0 mm after start of study treatment Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: Baseline and 12, 24, 48, 72, 96, 168 (192) hours after initiating treatment
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants
  48-72h | 2 | 0
  72-96h | 10 | 0
  96-192h | 45 | 10
  Not achieved | 41 | 92

7. Secondary Outcome: Responder Rate 1
Description: defined as the percentage of patients achieving ≥50% reduction from baseline in the VAS score for POM at 72 hours Visual Analogue Scale (VAS) 0 = "no pain", 100 = "Extreme pain"
Time Frame: 72 hours
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants | 93 | 15

8. Secondary Outcome: Global Efficacy Assessments 1 by Patient
Description: The global efficacy was assessed by the patients. The patients answered question below;
  -Considering all the ways this treatment has affected you since you started the clinical trial, how well are you doing? (5-point Likert scale: 0 = very good, 1 = good, 2 = fair, 3 = poor, and 4 = very poor). [Global efficacy assessment 1]
Time Frame: 48 h, 72 h, and 168 h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants
  48h: Very poor | 0 | 2
  48h: Poor | 0 | 13
  48h: Fair | 15 | 49
  48h: Good | 47 | 30
  48h: Very good | 36 | 8
  72h: Very poor | 0 | 1
  72h: Poor | 0 | 13
  72h: Fair | 6 | 46
  72h: Good | 41 | 31
  72h: Very good | 51 | 11
  168h: Very poor | 0 | 1
  168h: Poor | 0 | 11
  168h: Fair | 3 | 42
  168h: Good | 36 | 31
  168h: Very good | 59 | 17

9. Secondary Outcome: Global Efficacy Assessments 2 by Patient
Description: The global efficacy was assessed by the patients. The patients answered question below
  -How do you rate this medication as treatment for your soft injury/contusion? (5-point Likert scale: 0 = excellent, 1 = very good, 2 = good, 3 = fair, and 4 = poor). [Global efficacy assessment 2]
Time Frame: 48 h, 72 h, and 168 h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants
  48h: Poor | 0 | 11
  48h: Fair | 12 | 35
  48h: Good | 28 | 36
  48h: Very good | 47 | 15
  48h: Excellent | 11 | 5
  72h: Poor | 0 | 13
  72h: Fair | 7 | 36
  72h: Good | 27 | 32
  72h: Very good | 50 | 12
  72h: Excellent | 14 | 9
  168h: Poor | 0 | 12
  168h: Fair | 7 | 29
  168h: Good | 24 | 37
  168h: Very good | 46 | 13
  168h: Excellent | 21 | 11

10. Secondary Outcome: Global Efficacy Assessments 1 by Investigator
Description: The global efficacy was assessed by the investigator.
  -Considering all the ways this treatment has affected you since you started the clinical trial, how well are you doing? (5-point Likert scale: 0 = very good, 1 = good, 2 = fair, 3 = poor, and 4 = very poor). [Global efficacy assessment 1]
Time Frame: 48 h, 72 h, and 168 h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants
  48h: Very poor | 0 | 1
  48h: Poor | 1 | 20
  48h: Fair | 15 | 45
  48h: Good | 35 | 17
  48h: Very good | 47 | 19
  72h: Very poor | 0 | 0
  72h: Poor | 0 | 22
  72h: Fair | 8 | 46
  72h: Good | 35 | 14
  72h: Very good | 55 | 20
  168h: Very poor | 0 | 1
  168h: Poor | 0 | 19
  168h: Fair | 8 | 42
  168h: Good | 31 | 19
  168h: Very good | 59 | 21

11. Secondary Outcome: Use of Rescue Medication
Description: Rescue medication (paracetamol, 500 mg tablets, up to 3000 mg daily) was allowed during the study, except for the 6 hours prior to V5 (72 h).
Time Frame: 0-168h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants | 0 | 0

12. Secondary Outcome: Resolution of Soft Tissue Injury/Contusion
Description: Resolution of soft tissue injury/contusion was assessed by the Investigator at Visit 7 (168h).
Time Frame: 168h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants | 92 | 49

13. Secondary Outcome: SPID of POM VAS Changes
Description: The sum of pain intensity difference (SPID) of POM on VAS changes over 0-24 h, 0-48 h, 0-72 h, and 0-96 h were calculated.
  SPID was calculated as the area under the curve of the VAS difference from baseline value.
Time Frame: 0-24 h, 0-48 h, 0-72 h, and 0-96 h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Mean (Full Range); unit: SPID of POM on VAS (mm x h)
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
SPID of POM on VAS (mm x h)
  0-24 h | 342.5 [-36 to 1003] | 126.6 [-86 to 518]
  0-48 h | 1211.1 [423 to 2346] | 445.9 [-75 to 1614]
  0-72 h | 2425.1 [1133 to 4122] | 965.5 [-51 to 2982]
  0-96 h | 3881.4 [2156 to 5970] | 1753.7 [21 to 4178]

14. Secondary Outcome: Responder Rate 2 at 168h
Description: defined as the percentage of patients able to resume training/normal physical activity by 168 hours
Time Frame: 168h
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants | 92 | 49

15. Other Pre Specified Outcome: Adhesive Power of the Patch
Description: Adhesive power of the patch measured by a 5 point numerical scale (0= ≥ 90 % adhered, 1= ≥ 75 % to < 90 % adhered, 2= ≥ 50 % to < 75 % adhered, 3= > 0 % to <50 % adhered, 4=completely detached) at every visit except V1.
Time Frame: 12h for day 1, 24h for day 1-5 and 7 after application of each patch
Population: The Full Analysis Set (all randomized patients who received at least one dose of study drug).
Measure: Count of Units; unit: Number of patches
Units Other Than Participants: Number of patches
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Number analyzed (Number of patches) | 490 | 510
Number of patches
  12h: number analyzed (Number of patches) | 98 | 102
  12h: Completely detached | 1 | 0
  12h: ≥ 0 % to < 50 % adhered | 0 | 4
  12h: ≥ 50 % to < 75 % adhered | 23 | 27
  12h: ≥ 75 % to < 90 % adhered | 46 | 51
  12h: ≥ 90 % adhered | 28 | 20
  24h: Completely detached | 0 | 1
  24h: ≥ 0 % to < 50 % adhered | 10 | 10
  24h: ≥ 50 % to < 75 % adhered | 101 | 145
  24h: ≥ 75 % to < 90 % adhered | 202 | 206
  24h: ≥ 90 % adhered | 177 | 148

16. Other Pre Specified Outcome: Local Tolerability
Description: Local tolerability was assessed by the Investigator according to the following numerical scale:
  0: No evidence of irritation
  1. Minimal erythema, barely perceptible
  2. Definite erythema, readily visible, minimal edema or minimal papular response
  3. Erythema and papules
  4. Definite edema
  5. Erythema, edema and papules
  6. Vesicular eruption
  7. Strong reaction spreading beyond test site
Time Frame: 24, 48, 72, 96, 168h
Population: Safety Set (SAF) The safety set included all randomized patients who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Control Drug
Number analyzed (Participants) | 98 | 102
Participants
  24h: Minimal erythema (1) | 3 | 4
  24h: No evidence of irritation (0) | 95 | 98
  48h: Minimal erythema (1) | 3 | 9
  48h: No evidence of irritation (0) | 95 | 93
  72h: Minimal erythema (1) | 4 | 6
  72h: No evidence of irritation (0) | 94 | 96
  96h: Minimal erythema (1) | 1 | 4
  96h: No evidence of irritation (0) | 97 | 98
  168h: Minimal erythema (1) | 4 | 4
  168h: No evidence of irritation (0) | 94 | 98

ADVERSE EVENTS:
Time Frame: From Baseline assessment for up to 7 days (±1 days)
Arm/Group | Active Arm | Control Drug
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/102
Other Adverse Events (participants affected / at risk) | 9/98 | 16/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm (N=98) | Control Drug (N=102)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 8 (15) | 15 (27) — Observed at application site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT04908748/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT04908748/SAP_001.pdf